CLINICAL TRIAL: NCT00919542
Title: A Pilot (Double Blind Controlled) Study Randomizing Patients With New Acute ENL to Treatment Either With Ciclosporin or Prednisolone.
Brief Title: Ciclosporin in the Management of New Erythema Nodosum Leprosum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Homes and Hospitals of St Giles (Other); Alert Hospital, Ethiopia (Other); Armauer Hansen Research Institute, Ethiopia (Other)
Responsible Party: Principal Investigator, Saba Lambert, Clinical Research Fellow, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITCRBY24-ENLA
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Leprosy
Keywords: Leprosy; ENL; Erythema Nodosum Leprosum; Prednisolone; Ciclosporin
MeSH Terms: conditions — Leprosy | interventions — Cyclosporine; Prednisolone; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prednisolone (Active Comparator): standard course of prednisolone given in a reducing regimen over 16 weeks
  Interventions: Drug: prednisolone
- Ciclosporin (Experimental): ciclosporin reducing regimen lasting 16 weeks (additional prednisolone given for the first four weeks)
  Interventions: Drug: Ciclosporin

INTERVENTIONS:
Drug: Ciclosporin — Ciclosporin 7.5mg/kg - reducing regimen over 16 weeks (additional prednisolone given for the first four weeks)
  Other Names: cyclosporin; Cyclosporin A
  Arms: Ciclosporin
Drug: prednisolone — prednisolone 40mg daily then reducing regimen over 16 weeks
  Other Names: corticosteroids
  Arms: prednisolone

SUMMARY:
Study 2A: Ciclosporin in the management of new Erythema Nodosum Leprosum

Objective: A pilot (double blind controlled) study randomizing patients to treatment either with Ciclosporin or Prednisolone to assess the safety, tolerability and efficacy of Ciclosporin in the treatment of patients with new acute Type 2 reactions (ENL).

DETAILED DESCRIPTION:
A pilot (double blind controlled) study randomizing patients to treatment either with Ciclosporin or Prednisolone to assess the safety, tolerability and efficacy of Ciclosporin in the treatment of patients with new acute Type 2 reactions (ENL).

ELIGIBILITY:
Inclusion Criteria:

* Individuals with clinical evidence of new ENL
* Aged 18-65
* Weigh more than 30Kg

Exclusion Criteria:

* Unwillingness to give informed consent
* Patients with severe active infections such as tuberculosis
* Pregnant or breastfeeding women (see Appendix II)
* Those with renal failure, abnormal renal function, hypertensive
* Patients taking thalidomide currently or within the last 3 months
* Patients not willing to return for follow-up
* Women of reproductive age not willing to use contraception for the duration of the study ( see Appendix II)
* HIV positive patients

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Number of ENL recurrence episodes per patient | up to 32 weeks

SECONDARY OUTCOMES:
Mean time to ENL recurrence after initial control | up to 32 weeks
Amount of additional prednisolone required by patients | up to 32 weeks
Frequency of adverse events for patients in each treatment arm | up to 32 weeks
Difference in score in Quality of Life assessment between start and end for patients in each treatment arm | up to 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diana NJ Lockwood, MBchB, Study Director — London SHTM
Locations (1):
- Alert Hospital, Addis Ababa, Ethiopia